CLINICAL TRIAL: NCT05130424
Title: A Real-world Study of Herombopag in the Treatment of Thrombocytopenia Related Diseases in Henan Province
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SuxiaLuo (Other Government)
Responsible Party: Sponsor-Investigator, SuxiaLuo, chief physician, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Other Study IDs: HNHQRWS
Record Dates: First submitted 2021-10-28; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Carcinoma;Blood
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Herombopag — Herombopag in the treatment of thrombocytopenia-related diseases Non-interventional clinical research.Do not interfere with the dosage and market of Hetrobopar Oral medication

SUMMARY:
To observe and evaluate the safety and effectiveness of herombopag in the treatment of thrombocytopenia-related diseases in Henan Province

DETAILED DESCRIPTION:
This study is designed as a real-world study on the treatment of thrombocytopenia-related diseases with Herombopag, to observe and analyze the safety and efficacy of Herombopag for thrombocytopenia-related diseases in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Thrombocytopenia related diseases;
2. Volunteer to join this study and sign an informed consent form;
3. Clinical evaluation can benefit from Herombopag.

Exclusion Criteria:

1. Those who have been confirmed to be allergic to Herombopag and/or its excipients;
2. Pregnant or breastfeeding women;
3. Except for patients with contraindications to Herombopag;
4. Doctors evaluate patients who are not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thrombocytopenia-related diseases
Sampling Method: Non-Probability Sample
Enrollment: 498 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events after the treatment of Herombopag | From the treatment of Herombopag to 28 days after the end of the medication
  The investigator will observe incidence of adverse events after the treatment of Herombopag, including thrombosis, diarrhea, abnormal liver function and so on.

SECONDARY OUTCOMES:
Changes of the platelet counts after the treatment of Herombopag | From the treatment of Herombopag to 28 days after the end of the medication
  The investigator will assess the changes of the platelet counts after the treatment of Herombopag。
Proportion of patients with platelet transfusion | From the treatment of Herombopag to 28 days after the end of the medication
  The investigator will assess the proportion of patients with platelet transfusion after the treatment of Herombopag。

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China